CLINICAL TRIAL: NCT05164614
Title: A Phase I Study to Evaluate the Pharmacokinetics of Parathyroid Hormone (1-34) Administered Orally Via RaniPill™ Capsule
Brief Title: Study Evaluating PK of PTH Administered Orally Via RaniPill™ Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RANI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-0004
Record Dates: First submitted 2021-12-01; First posted 2021-12-20 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Forteo; Parathyroid Hormone; PTH
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Intervention Model Description: Healthy women volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RT-102 Group 1 (Experimental): In 15 subjects, a RaniPill capsule containing 20 µg of PTH will be administered and serial blood samples will be collected for PK analysis.
  Interventions: Combination Product: RT-102 (20 μg)
- RT-102 Group 2 (Experimental): In 15 subjects, a RaniPill capsule containing 80 µg of PTH will be administered and serial blood samples will be collected for PK analysis.
  Interventions: Combination Product: RT-102 (80 μg)
- SC Group (Active Comparator): In 10 subjects, 20 µg of Forteo will be administered subcutaneously and serial blood samples will be collected for PK analysis.
  Interventions: Drug: Forteo
- Part 2; Group 1 (Experimental): In up to 7 subjects, once-a-day repeat dosing with RT-102 (20 mcg) for 7 days in healthy post-menopausal or surgically sterile with bilateral oophorectomy women.
  Interventions: Combination Product: RT-102 (20 μg)
- Part 2; Group 2 (Experimental): In up to 12 subjects, once-a-day repeat dosing with RT-102 (20 mcg) for 7 days in healthy women.
  Interventions: Combination Product: RT-102 (20 μg)

INTERVENTIONS:
Combination Product: RT-102 (80 μg) — RaniPill capsule containing PTH with doses of 20 and 80 μg
  Arms: RT-102 Group 2
Drug: Forteo — A commercial formulation of PTH for SC control (20 µg)
  Arms: SC Group
Combination Product: RT-102 (20 μg) — RaniPill capsule containing PTH with dose of 20μg
  Arms: Part 2; Group 1; Part 2; Group 2; RT-102 Group 1

SUMMARY:
A prospective, single-center, open-label, phase I study evaluating the pharmacokinetics (PK) of human parathyroid hormone (1-34) ("PTH") administered via the RaniPill™ capsule ("RT-102").

DETAILED DESCRIPTION:
The RaniPill device is a capsule-like ingestible device, which injects a microneedle containing a micro tablet (payload/drug) into the intestinal wall. This is a single-center, prospective, open-label, feasibility study being conducted in two parts.

Part 1: Healthy women volunteers, 18-65 years of age, of any race, recruited from the general population and assigned to one of the following groups:

RT-102:

* RT-102 Group 1: 20 µg (N=15)
* RT-102 Group 2: 80 µg (N=15)

Subcutaneous (SC):

• SC Group: 20 µg of Forteo (N=10)

Part 2: Healthy women, 18-65 years of age, or healthy post-menopausal or surgically sterile with bilateral oophorectomy women of any race, recruited from the general population will have once-a-day repeat dosing with 20 μg dose of RT-102 for 7 days (N= up to 12):

* Healthy women: N = up to 12
* Post-menopausal or surgically sterile volunteers: N = up to 7

ELIGIBILITY:
Inclusion Criteria:

Part 1

1. Participant understands and voluntarily signs the approved informed consent document prior to the performance of any study-specific procedures
2. Willing to comply with all study procedures and available for the entire duration of the study
3. Participant is ambulatory female between 18 to 65 years of age.
4. BMI between 19 to 32 kg/m2.
5. In good health, determined by no clinically significant findings from medical history, physical examination, laboratory tests, and vital signs.
6. Non-menstruating, non-pregnant or non-lactating women during study participation NOTE: Females who are of childbearing potential must have had a negative pregnancy test on day of screening. Contraception (double barrier contraception and be protected by a daily combination birth control pill containing estrogen and progestin or any other form of hormonal contraceptive if cannot use the contraceptive pill) should be used between Screening visit and 30 days after dosing if actively engaged in penile-vaginal intercourse.

Part 2: Healthy Women

1. Participant understands and voluntarily signs the approved informed consent document prior to the performance of any study-specific procedures
2. Willing to comply with all study procedures and available for the entire duration of the study
3. Participant is ambulatory female between 18 to 65 years of age.
4. BMI between 19 to 32 kg/m2.
5. In good health, determined by no clinically significant findings from medical history, physical examination, laboratory tests, and vital signs.
6. Non-menstruating, non-pregnant or non-lactating women during study participation NOTE: Females who are of childbearing potential must have had a negative pregnancy test on day of screening. A double barrier approach using highly effective methods of contraception (e.g., oral contraceptives containing combined estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system [e.g., Mirena], progestogen-only hormonal contraception associated with inhibition of ovulation, nonhormonal intrauterine device, bilateral tubal occlusion) should be used between Screening visit and 30 days after dosing if actively engaged in penile-vaginal intercourse.

Part 2: Post-menopausal/surgically sterile

1. Participant understands and voluntarily signs the approved informed consent document prior to the performance of any study-specific procedures
2. Willing to comply with all study procedures and available for the entire duration of the study
3. Healthy ambulatory female post-menopausal for at least 1 year or surgically sterile with bilateral oophorectomy
4. BMI between 19 to 32 kg/m2.
5. In good health, determined by no clinically significant findings from medical history, physical examination, laboratory tests, and vital signs.

Exclusion Criteria:

Part 1

1. Participants with known history of chronic constipation, gastroparesis / delayed gastric emptying, gastric or duodenal ulcers, dysphagia, dyspepsia, esophagitis, esophageal spasm, GERD, IBD, Crohn's disease, stomas, tumors, ischemic or ulcerative colitis
2. Participant has known history of intolerance of PTH (1-34)
3. Participant has known history of high levels of uric acid outside normal ranges
4. Participant has known history of osteoporosis or other bone disorders (such as Paget's disease)
5. Participant has known history of Cushing's disease, hypo- or hyper-parathyroidism or malabsorptive syndromes within the past year
6. Participant is taking calcium and/or vitamin D supplements within 7 days of treatment (including multi-vitamins containing calcium and/or vitamin D)
7. Participant has febrile illness within 30 days of the study procedures
8. Participant currently treated with parathyroid hormone, parathyroid hormone-related peptide-derived drugs, or bone anabolic steroids, including abaloparatide, teriparatide, or parathyroid hormone (1-84)
9. Participant currently treated with intravenous bisphosphonates for at least 1 month or oral bisphosphonates within the past year (12 months). Subjects who have received a short course of oral bisphosphonate therapy (3 months or less) may be enrolled if the treatment occurred 6 or more months prior to enrollment
10. Participants on a regimen of proton pump inhibitors (e.g. omeprazole) or histamine H2 receptor antagonists (e.g. ranitidine)
11. Participants with known bowel obstruction/stricture/fistula
12. Participants who have undergone gastrointestinal surgery (Roux-en-Y, Billroth II, Whipple, intestinal resection for any reason)
13. Participants who have undergone a recent (less than a month) barium X-ray procedure
14. Participants with known allergies or sensitivity to contrast media or barium sulfate
15. Participant with history of chronic disease that in the investigator's judgement may impact subject safety or study outcomes
16. Participants with congestive heart failure, renal failure
17. Presence of cardiac pacemaker or implanted electromedical device
18. Participant who is pregnant or lactating
19. Participant has received an investigational or marketed drug during a trial within the past 1 month or 5 half-lives of the investigational drug, whichever is longer
20. Participant received COVID-19 vaccine within 7 days of dosing
21. Participant is unlikely, in the investigator's judgment, to be able to complete participation in the study as required per study plan
22. Any other history which, in the investigator's judgment, makes the participant ineligible or places the participant at risk

Part 2: Healthy Women

1. Participants with known history of chronic constipation, gastroparesis / delayed gastric emptying, gastric or duodenal ulcers, dysphagia, dyspepsia, esophagitis, esophageal spasm, GERD, IBD, Crohn's disease, stomas, tumors, ischemic or ulcerative colitis
2. Participant has known history of intolerance of PTH (1-34)
3. Participant has known history of high levels of uric acid outside normal ranges
4. Participant has known history of osteoporosis or other bone disorders (such as Paget's disease)
5. Participant has known history of Cushing's disease, hypo- or hyper-parathyroidism or malabsorptive syndromes within the past year
6. Participant is taking calcium and/or vitamin D supplements within 7 days of treatment (including multi-vitamins containing calcium and/or vitamin D)
7. Participant has febrile illness within 30 days of the study procedures
8. Participant currently treated with parathyroid hormone, parathyroid hormone-related peptide-derived drugs, or bone anabolic steroids, including abaloparatide, teriparatide, or parathyroid hormone (1-84)
9. Participant currently treated with intravenous bisphosphonates for at least 1 month or oral bisphosphonates within the past year (12 months). Subjects who have received a short course of oral bisphosphonate therapy (3 months or less) may be enrolled if the treatment occurred 6 or more months prior to enrollment
10. Participants on a higher than the lowest approved therapeutic dose regimen of proton pump inhibitors (see Section 8.3.9 for details)
11. Participants on a H2 receptor antagonists (e.g. ranitidine)
12. Participants with known bowel obstruction/stricture/fistula
13. Participants who have undergone gastrointestinal surgery (Roux-en-Y, Billroth II, Whipple, intestinal resection for any reason)
14. Participants who have undergone a recent (less than a month) barium X-ray procedure
15. Participants with known allergies or sensitivity to contrast media or barium sulfate
16. Participant with history of chronic disease that in the investigator's judgement may impact subject safety or study outcomes
17. Participants with congestive heart failure, renal failure
18. Presence of cardiac pacemaker or implanted electromedical device
19. Participant who is pregnant or lactating
20. Participant has received an investigational or marketed drug during a trial within the past 1 month or 5 half-lives of the investigational drug, whichever is longer
21. Participant received COVID-19 vaccine within 7 days of dosing
22. Participant is unlikely, in the investigator's judgment, to be able to complete participation in the study as required per study plan
23. Any other history which, in the investigator's judgment, makes the participant ineligible or places the participant at risk

Part 2: Post-menopausal/surgically sterile

1. Participants with known history of chronic constipation, gastroparesis / delayed gastric emptying, gastric or duodenal ulcers, dysphagia, dyspepsia, esophagitis, esophageal spasm, GERD, IBD, Crohn's disease, stomas, tumors, ischemic or ulcerative colitis
2. Participant has known history of intolerance of PTH (1-34)
3. Participant has known history of high levels of uric acid outside normal ranges
4. Participant has known history of osteoporosis or other bone disorders (such as Paget's disease)
5. Participant has known history of Cushing's disease, hypo- or hyper-parathyroidism or malabsorptive syndromes within the past year
6. Participant is taking calcium and/or vitamin D supplements within 7 days of treatment (including multi-vitamins containing calcium and/or vitamin D)
7. Participant has febrile illness within 30 days of the study procedures
8. Participant currently treated with parathyroid hormone, parathyroid hormone-related peptide-derived drugs, or bone anabolic steroids, including abaloparatide, teriparatide, or parathyroid hormone (1-84)
9. Participant currently treated with intravenous bisphosphonates for at least 1 month or oral bisphosphonates within the past year (12 months). Subjects who have received a short course of oral bisphosphonate therapy (3 months or less) may be enrolled if the treatment occurred 6 or more months prior to enrollment
10. Participants on a higher than the lowest approved therapeutic dose regimen of proton pump inhibitors (see Section 8.3.9 for details)
11. Participants on a H2 receptor antagonists (e.g. ranitidine)
12. Participants with known bowel obstruction/stricture/fistula
13. Participants who have undergone gastrointestinal surgery (Roux-en-Y, Billroth II, Whipple, intestinal resection for any reason)
14. Participants who have undergone a recent (less than a month) barium X-ray procedure
15. Participants with known allergies or sensitivity to contrast media or barium sulfate
16. Participant with history of chronic disease that in the investigator's judgement may impact subject safety or study outcomes
17. Participants with congestive heart failure, renal failure
18. Presence of cardiac pacemaker or implanted electromedical device
19. Participant has received an investigational or marketed drug during a trial within the past 1 month or 5 half-lives of the investigational drug, whichever is longer
20. Participant received COVID-19 vaccine within 7 days of dosing
21. Participant is unlikely, in the investigator's judgment, to be able to complete participation in the study as required per study plan
22. Any other history which, in the investigator's judgment, makes the participant ineligible or places the participant at risk

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Evaluate Cmax of PTH administered via the RaniPill capsule | Within 24 hours after ingestion of the device
  To obtain PK profiles of single doses of PTH given via RaniPill™ capsule in healthy participants with doses of 20 and 80 μg. Cmax of PTH will be calculated from the PK profiles.
Evaluate Tmax of PTH administered via the RaniPill capsule | Within 24 hours after ingestion of the device
  To obtain PK profiles of single doses of PTH given via RaniPill™ capsule in healthy participants with doses of 20 and 80 μg. Tmax of PTH will be calculated from the PK profiles.
Evaluate AUC of PTH administered via the RaniPill capsule | Within 24 hours after ingestion of the device
  To obtain PK profiles of single doses of PTH given via RaniPill™ capsule in healthy participants with doses of 20 and 80 μg. Absorption (AUC) of PTH will be calculated from the PK profiles.

SECONDARY OUTCOMES:
Safety and tolerability of RT-102 | Within 24 hours after ingestion of the device
  Monitoring and recording of adverse events possibly related to RT-102.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Myers, Study Director — RANI Therapeutics
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No